CLINICAL TRIAL: NCT00400933
Title: Evaluation of a Six-session Psycho-education Group Program Delivered to Family Members and Close Friends of Patients Suffering From Eating Disorders and Co-morbid Personality Disorders
Brief Title: Evaluation of a Six-session Psycho-education Group Program
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: shortage of experienced health care personnel after reorganisation of units
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 4,2006.2005
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Eating Disorders; Personality Disorders
Keywords: Psycho-education; Eating disorders; Personality disorders; Relatives and close friends; Caregiver burden
MeSH Terms: conditions — Feeding and Eating Disorders; Personality Disorders; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- psycho-education (Experimental): six session psycho-educational group program for family members and close friends of persons with eating disorders and co-morbid personality disorders
  Interventions: Behavioral: psycho-education

INTERVENTIONS:
Behavioral: psycho-education — six session psycho-educational group program for family members and close friends of persons with eating disorders and co-morbid personality disorders

SUMMARY:
The aim of this project is to analyze the impact of a psycho-educational group program on the family members and close friends of persons with eating disorders and co-morbid personality disorders.

DETAILED DESCRIPTION:
The aim of this project is to analyze the impact of a six session psycho-educational group program on the family members and close friends of persons with eating disorders and co-morbid personality disorders.

Measurements: General health, perceived caregiver burden, and relation to the patient at the following point of time: pre -, post- and follow up, with waiting list control.

ELIGIBILITY:
Inclusion Criteria:

* Relatives and close friends to persons receiving treatment for their eating disorder and comorbid personality disorder.
* > 18 years,
* Speak and understand norwegian language, and
* Informed consent to participate for both relative and patient.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-11; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Scores on perceived caregiver burden (Experience of Caregiving Inventory [ECI]) | 1 year

SECONDARY OUTCOMES:
Scores on general health and relational variables | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Are Holen, PhD MD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Østmarka Psychiatric Department, St Olavs Hospital, University Hospital of Trondheim, Trondheim, Trondheim, Norway